CLINICAL TRIAL: NCT06909721
Title: Misoprostol Versus Dinoprostone in Induction of Labor,Randomized Controlled Study
Brief Title: Misoprostol Versus Dinoprostone in Induction of Labor
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Shaimaa Elkhodary Hassan, Resident of Obstetrics & Gynecology, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Shaimaa Elkhodary
Record Dates: First submitted 2025-03-19; First posted 2025-04-03 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2023-06

CONDITIONS: Induction of Labor
MeSH Terms: interventions — Misoprostol; Dinoprostone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Misoprostol Group (Active Comparator): About 100 pregnant women received Misoprostol vaginal tablets (25-50 mcg every 6 Hours for 4 doeses and re use after 48 hour) for induction of normal labour
  Interventions: Drug: Misoprostol
- Dinoprostone Group (Active Comparator): About 100 pregnant women received Dinoprostone vaginal tablets (3mg vaginal tablets, one tablet to be inserted high in posterior fornix and the second tablet inserted after 8 hour if labour not established with maximum does 6 mg) for induction of normal labour
  Interventions: Drug: Misoprostol

INTERVENTIONS:
Drug: Misoprostol — to compare Misoprostol and Dinoprostone as regarding to cost-effectiveness and safety in induction of normal Labor
  Other Names: Dinoprostone

SUMMARY:
Endogenous prostaglandins, derived from the uterus, cervix, placenta, and membranes of fetus, are essential for cervical ripening ,the investigators aimed to compare Misoprostol and Dinoprostone as regarding to cost-effectiveness and safety in induction of Labor.

Both misoprostol and dinoprostone have demonstrated efficiently in cervical ripening and labor induction. However, their use must be carefully monitored to minimize risks and optimize outcomes. Factors such as parity, gestational age, maternal medical history, and the indication for induction should be considered when selecting the most appropriate induction method. Additionally, patient preferences and institutional protocols play a role in decision-making.

Recent advancements in IOL techniques include the use of combination methods, like mechanical and pharmacological agents, to enhance efficacy and reduce complications. For example, the combination of a Foley catheter with low-dose misoprostol has been shown to improve cervical ripening and reduce the time to delivery . Additionally, the development of new pharmacological agents, such as misoprostol vaginal inserts and controlled-release dinoprostone gels, offers promising alternatives for safe and effective labor induction.

DETAILED DESCRIPTION:
Induction of labor (IOL) is a critical obstetric technique utilized to trigger uterine contractions artificially after fetal viability but prior to the spontaneous onset of labor. It is primarily aimed at achieving cervical effacement and dilatation to facilitate vaginal delivery. This intervention is often necessary in various clinical scenarios, like post-term pregnancies, preeclampsia, gestational diabetes, intrauterine growth restriction, or maternal medical conditions that pose risks to the mother or fetus. Globally, IOL is performed in up to 25% of pregnancies, highlighting its importance in modern obstetrics . In Europe, the rates of IOL vary significantly, ranging from 7% to 33%, reflecting differences in healthcare systems, clinical guidelines, and patient demographics .

The success of IOL is heavily influenced by the condition of cervix at the time of induction. Cervical status is assessed using the Bishop's scoring system, which evaluates factors like cervical dilatation, effacement, consistency, position, and fetal station. A favorable cervix, characterized by a Bishop's score of 6 or higher, is related to an elevated probability of successful vaginal delivery. In contrast, an unfavorable cervix (posterior, firm, and long) presents significant challenges, decreasing the chances of vaginal birth and increasing the risk of cesarean delivery.

Cervical ripening is a fundamental process that prepares the cervix for labor by increasing its softness and distensibility. This process is controlled by a complex interplay of hormonal, biochemical, vasodilatory and inflammatory alterations. Endogenous prostaglandins (PGs), produced by uterus, cervix, fetal membranes and placenta, have a pivotal role in these changes. PGs stimulate the breakdown of collagen fibers, increase water content, and promote the release of cytokines and other inflammatory mediators that facilitate cervical remodeling. When natural ripening is insufficient, iatrogenic methods are employed to induce cervical ripening and labor. These methods include mechanical agents, such as Foley catheters, cervical dilators, or amniotomy, and pharmacological agents, such as prostaglandins, oxytocin, and smooth muscle stimulants like herbs or castor oil.

Despite its widespread use, IOL is not without risks. Common challenges include ineffective labor induction, prolonged labor, and excessive uterine activity, which may result in complications like fetal distress, uterine rupture, and an elevated probability of cesarean delivery. Prostaglandins, which mediate their effects through specific G protein-coupled receptors (GPCRs), are integral to the inflammatory and immune responses that drive cervical ripening .

However, the therapeutic utilization of natural PGs is restricted by their quick metabolism, chemical instability, and short half-life, as well as their propensity to cause side effects like vomiting, diarrhea, nausea, and uterine hyperstimulation .

To overcome these limitations, synthetic prostaglandins have been developed and are widely used in clinical practice. Misoprostol, a synthetic analog of prostaglandin E1 (PGE1), is the most frequently utilized agent due to its stability, cost-effectiveness, and ease of administration. It is available in oral, sublingual, and vaginal forms, making it a versatile option for labor induction. Misoprostol is particularly effective in low-resource settings because of its affordability and stability at room temperature. However, its use requires careful dosing to avoid complications such as uterine hyperstimulation and fetal distress .

Dinoprostone, a synthetic analog of prostaglandin E2 (PGE2), is another widely used agent, particularly in settings where controlled release and fewer side effects are desired. Dinoprostone is available in gel, insert, and suppository forms, allowing for tailored dosing based on individual patient needs. It is often preferred in cases where a slower, more controlled induction process is warranted. However, dinoprostone is more expensive than misoprostol and requires refrigeration, which can limit its use in resource-constrained settings.

ELIGIBILITY:
Inclusion Criteria:

* Singleton pregnancy
* Intact membranes
* Bishop score 4-6 or less
* Women accepted to participate in the study
* Indicated patient of induction 39WeeKs of pregnancy or more

Exclusion Criteria:

* Fetal congenital anomalies
* malpresentation
* irregular fetal heart rate patterns
* placental abnormalities, and any contraindications to administering prostaglandins
* involving a history of glaucoma, asthma, cardiovascular disease or preexisting cardiac
* prior uterine operation, cesarean delivery
* maternal chronic illness

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Actual)
Dates: Start 2023-06-10 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-06-10 (Actual)

PRIMARY OUTCOMES:
Induction of Labor | 48 hours after drug administration
  Assessment of labour induction by the using the modified Bishop score . The bishop score evaluated cervical readiness for labor induction by examining five components: cervical consistency, cervical dilation, station of the baby, cervical position, and cervical length. Cervical dilation measured the opening of the cervix on a scale from 0 (no dilation) to 3 (≥5 cm). Cervical consistency assessed the texture of the cervix, scored from 0 (firm) to 2 (soft). Cervical position was rated from 0 (posterior) to 2 (anterior). The baby's station was scored from -3 (high in the pelvis) to +3 (deeply engaged). Cervical length was evaluated on a scale from 0 (≥3 cm) to 2 (<2 cm). These components were combined to produce a total Bishop score varying from 0 to 13.
Induction of Labor | just after delivery
  Assessment of labour induction by the using the Apgar score. The Apgar score, performed at one and five minutes after birth, assessed the newborn's condition across five factors: respiratory effort, heart rate, reflex irritability, tone of muscle, and color of skin, with each scored from zero to two. Heart rate was rated as 2 if it exceeded 100 beats per minute, 1 if below 100, and 0 if absent.

CONTACTS AND LOCATIONS:
Overall Officials: Mahmoud Ebrahim Al Rashidi, Professor, Study Chair — Obstetrics and Gynecology Department, Faculty of medicine,Al-Azhar University, Assiut.
Locations (1):
- Al-Azhar University Hospitals, Asyut, Assuit, Egypt

IPD SHARING:
Plan to Share IPD: Undecided